CLINICAL TRIAL: NCT00087334
Title: A Phase I/II Study of Capecitabine (XELODA®, Roche) Plus Oxaliplatin (Eloxatin®, Sanofi) Plus ZD 1893 (IRESSA®) in the Treatment of Metastatic Colorectal Cancer
Brief Title: Capecitabine, Oxaliplatin, and Gefitinib in Treating Patients With Metastatic Colorectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to poor/low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: I 17403; RPCI-I-17403; ZENECA-IRUSIRES0414
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Gefitinib; Oxaliplatin

INTERVENTIONS:
Drug: capecitabine
Drug: gefitinib
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and oxaliplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Combining capecitabine and oxaliplatin with gefitinib may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of capecitabine when given together with oxaliplatin and gefitinib and to see how well they work in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of capecitabine when given in combination with oxaliplatin and gefitinib in patients with metastatic colorectal cancer. (phase I)
* Determine the response rate in patients treated with this regimen. (phase II)

Secondary

* Determine the safety and toxic effects of this regimen in these patients.
* Determine the 1-year survival of patients treated with this regimen. (phase II)
* Determine the progression-free and overall survival of patients treated with this regimen. (phase II)

OUTLINE: This is an open-label, nonrandomized, phase I, dose-escalation study of capecitabine followed by a phase II study.

* Phase I: Patients receive oral capecitabine twice daily on days 1-14 and oxaliplatin IV over 2 hours on day 1. Patients also receive oral gefitinib once daily beginning 5 days before the initiation of capecitabine and oxaliplatin and continuing for the duration of study treatment. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of capecitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II: Patients receive oral capecitabine (at the MTD determined in phase I), oxaliplatin IV, and oral gefitinib as in phase I.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 3-24 patients will be accrued for the phase I portion of this study within 1-12 months; and a total of 26 patients will be accrued for the phase II portion of this study within 8-13 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed* colorectal cancer

  * Metastatic disease
  * The site of the primary tumor must have been confirmed endoscopically, radiologically, or surgically to be the colon or rectum NOTE: *Confirmation is not required for recurrent metastatic disease unless an interval of > 5 years has elapsed between the initial primary surgery and the development of metastases
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 80

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL (transfusion allowed)

Hepatic

* AST and ALT ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ ULN
* No unstable or uncompensated hepatic disease

Renal

* Creatinine < 1.5 times ULN OR
* Creatinine clearance > 60 mL/min
* No unstable or uncompensated renal disease

Cardiovascular

* No unstable or uncompensated cardiac disease

Pulmonary

* No evidence of clinically active interstitial lung disease

  * Asymptomatic patients with chronic stable radiographic changes are eligible
* No unstable or uncompensated respiratory disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No known hypersensitivity to gefitinib or any of its excipients
* No known hypersensitivity to platinum compounds, fluorouracil, or capecitabine
* No severe or uncontrolled systemic disease
* Able to receive oral medication
* No known dihydropyrimidine dehydrogenase (DPD) deficiency
* No known peripheral neuropathy ≥ grade 1

  * Absence of deep tendon reflexes as the sole neurological abnormality allowed
* No other significant clinical disorder or laboratory finding that would preclude study participation
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix (phase II only)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* At least 4 weeks since prior chemotherapy for metastatic colorectal cancer (phase I)
* No prior chemotherapy for metastatic disease (phase II)

  * Prior fluorouracil and leucovorin calcium in the adjuvant setting allowed provided the last treatment was administered more than 6 months before the development of metastatic disease
* No prior irinotecan and oxaliplatin (phase II)

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent radiotherapy for colorectal cancer

Surgery

* See Disease Characteristics
* More than 4 weeks since prior major surgery (e.g., laparotomy)

Other

* Recovered from all prior therapy (no unresolved chronic toxicity > grade 2)
* More than 4 weeks since prior investigational drugs
* No prior epidermal growth factor receptor inhibitor therapy (phase II)
* No concurrent phenytoin, carbamazepine, rifampin, barbiturates, or Hypericum perforatum (St. John's wort)
* No other concurrent investigational drugs
* No other concurrent systemic therapy for colorectal cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-01; Primary Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose
Response rate

SECONDARY OUTCOMES:
Toxicity
1-year survival (phase II)
Progression-free survival (phase II)
Overall survival in (phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States